CLINICAL TRIAL: NCT04967833
Title: A Clinical Study to Evaluate the Safety and Efficacy of Autologous Tumor Infiltrating Lymphocytes Injection in Patients With Advanced Malignant Solid Tumors
Brief Title: A Study of GC101 TIL in Advanced Solid Tumors (TR)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Juncell Therapeutics (Industry)
Collaborators: Shanghai Tong Ren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC101-2021-TR-ST
Record Dates: First submitted 2021-06-10; First posted 2021-07-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors
Keywords: TIL,Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor Infiltrating Lymphocytes (Experimental): 1x10^9-5x10^10 in vitro expanded autologous TILs will be infused i.v. to patients with advanced solid tumors after NMA lymphodepletion treatment with hydroxychloroquine(600mg,single-dose) and cyclophosphamide.
  Interventions: Biological: Tumor Infiltrating Lymphocytes (TIL)

INTERVENTIONS:
Biological: Tumor Infiltrating Lymphocytes (TIL) — Biological: Tumor Infiltrating Lymphocytes (TIL) Adoptive transfer of 1x10^9-5x10^10 autologous TILs to patients i.v. in 30-120 minutes.

SUMMARY:
This study is to investigate the safety and efficacy of tumor infiltrating lymphocyte (TIL) therapy in patients with Advanced malignant solid tumors.Autologous TILs are expanded from tumor resections or biopsies and infused i.v. into the patient after NMA lymphodepletion treatment with hydroxychloroquine(600mg,single-dose) and cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years to 75 years;
2. Histologically diagnosed as primary/relapsed/metastasized malignant tumors;
3. Expected life-span more than 3 months;
4. Karnofsky≥60% or ECOG score 0-2;
5. Test subjects have failed standard treatment regimens, or there are no standard treatment regimens available.
6. Test subjects must have tumor regions eligible for biopsy or resection, or malignant body fluid where TILs can be isolated;
7. At least 1 evaluable tumor lesion;
8. Hematology and Chemistry（within 7 days prior to enrollment）:

   * Absolute count of white blood cells≥2.5×10^9/L;
   * Absolute count of neutropils≥1.5×10^9/L;
   * Absolute count of lymphocytes ≥0.7×109/L；
   * Platelet count≥100×10^9；
   * hemoglobin≥90 g/L;
   * Activated partial thromboplastin time (APTT) ≤1.5xULN (Unless received anticoagulant therapy within the previous 3 days);
   * International normalized ratio (INR) ≤1.5xULN (Unless received anticoagulant therapy within the previous 3 days);
   * Serum creatinine ≤1.5mg/dL(or ≤132.6μmol/L), or clearance rate≥50mL/min;
   * Serum ALT/AST ≤3×ULN(subjects with liver metastasis ≤3×ULN);
   * Totol bilirubin≤1.5×ULN;
9. No absolute or relative contraindications to operation or biopsy;
10. Test subjects with child-bearing potential must be willing to practice approved highly effective methods of contraception at the time of informed consent, and continue within 1 year after the completion of lymphodepletion；
11. Any malignant tumor-targeting therapies, including radiotherapy, chemotherapy and biologics must cease 28 days before obtaining TILs;
12. Be able to understand and sign the informed consent document;
13. Be able to stick to follow-up visit plan and other requirements in the agreement.

Exclusion Criteria:

1. Need glucocorticoid treatment, and daily dose of Prednisone greater than 15mg (or equivalent doses of hormones) or outoimmune diseases requiring immunomodulatory treatment;
2. Forced expiratory volume in one second (FEV1) less than 2L, diffusing capacity of the lung for carbon monoxide (DLCO) (calibrated) less than 40%;
3. Significant cardiovascular anomalies according to any of the following definition: New York Heart Association (NYHA) Grade III or IV congestive heart failure, clinically significant low blood pressure, uncontrollable symptomatic coronary artery diseases, or ejection fraction less than 35%; Severe cardiac rhythm and conduction anomaly, such as ventricular arrhythmia requiring clinical intervention, second-third degree atrio-ventricular conductive block, etc.
4. Human immunodeficiency virus (HIV) infection or anti-HIV antibody positive, active HBV or HCV infection (HBsAg positive and/or anti-HCV positive), syphilis infection or Treponema pallidum antibody positive;
5. Severe physical or mental diseases;
6. Have a systemic active infection requiring treatment, or have positive blood cultures(or imaging evidence of infection);
7. Having been treated within a month or being treated now with other medicines, or other biologic therapy, chemo-or radiotherapy;
8. History of allergy to chemical compound consisting of chemical and biologic substances resembling cell therapy;
9. Having received immunotherapy and developed irAE level greater than Level 3;
10. Previous anti-tumor treatment AE did not return to CTCAE5.0 version grade 1 or below (toxicity considered by the investigator as non-safety concerns like alopecia excluded);
11. Females in pregnancy or lactation;
12. History of organ transplantation, allogeneic stem cell transplantation, and renal replacement therapy;
13. Researchers considering the test subject as having a history of other severe systemic diseases, or other reasons inappropriate for the clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
Adverse Events(AE) | 6 month
  To characterize the safety profile of GC101 TIL in patients with recurrent, metastatic, or persistent solid tumor as assessed by incidence of adverse events.
Objective Response Rate (ORR) | Up to 36 months
  Proportion of patients with response per Response Evaluation Criteria in Solid Tumors (RECIST v1.1):
  ORR (proportion of patients) = # with CR + # with PR / # with CR + # with PR + # with SD + # with PD.
  ( Except baseline evaluation within 28 days before GC101 TIL infusion，PET/CT scan will be performed at 6 weeks after TIL infusion, and than every 6 weeks for 6 months, and then every 6 months after that for up to 3 years)

SECONDARY OUTCOMES:
Disease Control Rate (DCR） | Up to 36 months
  Percentage of patients that meet CR, PR and SD criteria set in this study according to RECIST v1.1： DCR (proportion of patients) = # with CR + # with PR + # with SD / # with CR + # with PR + # with SD + # with PD.
Duration of Response (DOR) | Up to 36 months
  The time length between the first confirmed objective response per RECIST 1.1 to the treatment and the subsequent disease progression per RECIST 1.1
Progression-Free Survival (PFS) | Up to 36 months
  The time length between GC101 TIL infusion and confirmed subsequent disease progression according to RECIST 1.1
Overall Survival (OS) | Up to 36 months
  The length of time from the date of the start of GC101-TIL treatment that the patients are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: LiJun Ma, Principal Investigator — Tongren Hospital,Shanghai Jiao Tong University School of Medicine
Locations (1):
- Tongren Hospital Shanghai Jiao Tong University School Of Medicine., Shanghai, China

IPD SHARING:
Plan to Share IPD: No